CLINICAL TRIAL: NCT06747910
Title: Assessment of Remote Approaches for Identification of Autonomic Dysfunction Among Survivors of Leukemia and Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: READ; NCI-2025-00603 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2024-12-12; First posted 2024-12-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Childhood Cancer
Keywords: Survivor; Acute lymphoblastic leukemia; Hodgkins's lymphoma; Autonomic
MeSH Terms: conditions — Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Physical Examination

STUDY DESIGN:
Intervention Model Description: Participants will complete an in-person assessment questionnaire for autonomic dysfunction (AD), during a scheduled on-campus SJLIFE visit and a remote assessment. Participants will be randomly assigned to either complete the AD symptom questionnaire before or after the standardized clinical AD assessment. Participants will be asked to wear a heart rate variability monitor for 7 days after the on-campus visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening (COMPASS31 + battery assessment + heart monitor) (Experimental): Patients complete the COMPASS31 questionnaire and undergo an in-person Ewing battery assessment over 60-90 minutes on study. Patients then wear a biosensensor heart monitor for 7 days to monitor heart rate variability remotely on study.
  Interventions: Other: Exercise Intervention - Ewing Battery Assessment; Other: Questionnaire Administration; Device: Medical Device Usage and Evaluation
- Screening (battery assessment + COMPASS31 + heart monitor) (Experimental): Patients undergo an in-person Ewing battery assessment over 60-90 minutes and complete the COMPASS31 questionnaire on study. Patients then wear a biosensensor heart monitor for 7 days to monitor heart rate variability remotely on study.
  Interventions: Other: Exercise Intervention - Ewing Battery Assessment; Other: Questionnaire Administration; Device: Medical Device Usage and Evaluation

INTERVENTIONS:
Other: Exercise Intervention - Ewing Battery Assessment — Undergo in-person Ewing battery assessment
Other: Questionnaire Administration — Receive COMPASS31 questionnaire
Device: Medical Device Usage and Evaluation — Wear biosensensor heart monitor that remotely collects heart rate variability.

SUMMARY:
This study seeks to determine if diagnosing cardiac autonomic dysfunction (AD) can be done remotely with the same accuracy as in-person testing. If so, the identification of AD could happen sooner, facilitating remote studies of the condition and potentially reducing the risk of illness. Childhood cancer survivors, particularly survivors of acute lymphoblastic leukemia (ALL) and Hodgkins's lymphoma (HL), appear to be at increased risk for AD.

Primary Objectives:

* To determine the sensitivity and specificity of heart rate variability (HRV), measured remotely with biosensor technology (Actigraph LEAP), compared to in-person assessment using the Ewing battery as the reference standard to identify cardiac autonomic dysfunction (AD) among survivors of leukemia and lymphoma.
* To determine the sensitivity and specificity of the Composite Autonomic Symptom Scale 31 (COMPASS31) compared to the Ewing battery to identify AD among leukemia and lymphoma survivors.

DETAILED DESCRIPTION:
Each participant will complete an in-person standardized clinical assessment for AD, called the Ewing battery. during the participants' Human Performance Lab during their SJLIFE functional exam. It is estimated it will take 60-90-minutes to complete the Ewing battery. The tests include monitoring heart rate variations during deep breathing and lying down to standing, as well as monitoring blood pressure variations when standing and maintaining hand grip. Participants will be asked to not consume aspirin, ibuprofen or acetaminophen 24-hours before the assessment. Additionally, participants will be asked to avoid alcohol or caffeine within 6-hours, and smoking 3-hours, before testing.

After the in-person assessment, each participant will be given a wrist biosensor to remotely monitor heart rate variability for 7 days after they return home. Participants will also complete an AD symptom questionnaire, COMPASS31. The AD symptom questionnaire will be completed either before or after the in-person assessment. This questionnaire will take about 20-30 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in St. Jude Lifetime Cohort (SJLIFE) >18 years of age.
* Primary diagnosis of acute lymphoblastic leukemia (ALL), Hodgkin's Lymphoma (HL), or Non-Hodgkin's Lymphoma (Non-HL).
* Not currently taking beta-blocker medication.

Exclusion Criteria:

* Individuals who cannot speak, read, and/or understand English.
* Individuals who are unable to follow directions/instructions in order to complete the Ewing battery.
* Individuals with acute heart failure (new or worsening signs and symptoms of heart failure, including a combination of the following: dyspnea, orthopnea, lower limb swelling, elevated jugular venous pressure, and pulmonary congestion).
* Women who are currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability (msec) | Up to 7 days after the on-campus study visit
  The standard deviation of normal-to-normal heartbeat intervals over a 24-hour period measured in milliseconds
Abbreviated Composite Autonomic Symptom Score (0-100) | During the on-campus study visit (Day 1)
  Symptom burden-based questionnaire of six weighted domains (orthostatic intolerance, vasomotor, secretomotor, gastrointestinal bladder and pupillomotor)
  Abbreviated Composite Autonomic Symptom Score:
  * This questionnaire, administered during Day 1, generates a weighted score from 0 to 100, and questions fall into one of six domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor function. Scores are determined by applying a simplified scoring algorithm.
  * Overall score interpretation:
    * < 3 or less: Mild
    * 3-7: Moderate
    * >7: Severe
Ewing Score (0-5) | During the on-campus study visit (Day 1)
  Derived from sum of five individual autonomic test scores
  Ewing Battery Scoring:
  * This battery is administered during Day 1. Each test within the battery (5 tests total) is assigned a score of 0 (normal), 0.5 (borderline), or 1 (abnormal).
  * Overall score interpretation:
    * 0-1: Considered normal autonomic function
    * 1.5-2: Mild autonomic dysfunction
    * 2.5-3: Moderate autonomic dysfunction
    * 3.5-5: Severe autonomic dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Wilson, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the ClinicalTrials.gov (CTG) website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols